CLINICAL TRIAL: NCT05289115
Title: Protocol for Assistance to Patients With Long Covid-19 Undergoing Treatment With HD-tDCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Suellen Marinho Andrade, Principal Investigator, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LongCOVID/HD-tDCS
Record Dates: First submitted 2022-03-16; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Coronavirus; COVID-19 Respiratory Infection
Keywords: COVID-19 Respiratory Infection; Transcranial direct current stimulation; Non-invasive brain stimulation; Electroencephalography; Long Covid
MeSH Terms: conditions — Coronavirus Infections; Post-Acute COVID-19 Syndrome | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental Group/ Active HD-tDCS (Experimental): Patients who will be randomly enrolled in this group. They will receive 10 sessions of anodal stimulation on cortical representation zone of left diaphragmatic motor cortex using HD-tDCS associated to respiratory training; for 20 minutes (each session) with a 3mA intensity. The electrical current will be delivered with a ramp-up time of 30 s, held at 3mA for 20 min, and then ramped down over 30 s.
  Interventions: Device: Experimental group/ Active HD-tDCS
- Control Group / Sham Group (Sham Comparator): Patients enrolled in this group condition will receive 10 sessions of anodal stimulation on cortical representation zone of left diaphragmatic motor cortex using HD-tDCS associated to respiratory training; for 20 minutes (each session) with a 3mA intensity. In the sham condition, the device will provide a 30-second ramp-up followed immediately by a 30-second ramp down.
  Interventions: Device: Control Group / Sham Group

INTERVENTIONS:
Device: Experimental group/ Active HD-tDCS — Patients enrolled in this group will received 20 minutes of anodal HD-tDCS ( tDCS 1x1, developed by Soterix Medical Inc.) during 10 sessions. It will be delivered a 3mA intensity electrical current accordingly 10/20 International System on cortical representation zone of left diaphragmatic motor cortex using HD-tDCS.
  Arms: Experimental Group/ Active HD-tDCS
Device: Control Group / Sham Group — 10-sessions of anodal HD-tDCS( tDCS 1x1, developed by Soterix Medical Inc.) associated to respiratory training; for 20 minutes (each session) with a 3mA intensity.The device will provide a 30-second ramp-up followed immediately by a 30-second ramp down.
  Arms: Control Group / Sham Group

SUMMARY:
COVID-19 is an infectious disease which presents a heterogenous clinical presentation. Recent investigations suggest that people who were infected by COVID-19 often develop physical disabilities (i.e. pain, fatigue) and neurological complications after hospital discharge. Many therapeutic approaches such as transcranial direct current stimulation high definition (HD-tDCS) have been proposed to minimize functional and structural impairments. Recently, I electroencephalogram (EEG) has been used as predictor of HD-tDCS effectiveness in diverse neurological populations. However, evidences about this tool utilization as efficacy predictor of tDCS in COVID-19 people rest inconclusive. Thereby, our objective is to evaluate HD-tDCS efficacy on fatigue, pain and functional capacity of patients with COVID-19 chronic.

DETAILED DESCRIPTION:
We propose a sham-controlled randomized clinical trial with patients in COVID-19 chronic. They will be evaluated according to following eligibility criteria :

Patients who had a medical diagnosis of COVID-19, clinically stable, able to respond to simple commands, able to walk for six minutes and who sign study consent form will be enrolled. Those who present associated neurological diseases, pregnant, users of psychoactive drugs, patients who have metallic implants, electronic devices, pacemakers, or epileptic patients will be excluded.

Patients will be allocated randomly to the experimental group or sham control. Sessions for experimental group consist of anodal HD-tDCS on Left diaphragmatic primary motor cortex associated to respiratory training (10 sessions, 3mA, 20 minutes/session). In the sham condition, the device provided a 30-second ramp-up period to the full 3 mA, followed immediately by a 30-second ramp down.

Patients will be assessed in three moments: pre-treatment, post-treatment and after 30 days treatment ending (follow-up).

ELIGIBILITY:
Patients who had a medical diagnosis of COVID-19, clinically stable, able to respond to simple commands, able to walk for six minutes and who sign study consent form will be enrolled. Those who present associated neurological diseases, pregnant, users of psychoactive drugs, patients who have metallic implants, electronic devices, pacemakers, or epileptic patients will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-04-14 (Estimated); Study Completion 2022-07-14 (Estimated)

PRIMARY OUTCOMES:
Fatigue Impact | From date of randomization (1 week before intervention beginning) up to 5 weeks (T1) and up to 10 weeks (T2; follow-up)
  MFIS-BR is a tool composed by 21 items stratified into 3 domains

SECONDARY OUTCOMES:
Pain Level | From date of randomization (1 week before intervention beginning) up to 5 weeks (T1) and up to 10 weeks (T2; follow-up)
  Pain level will be evaluated through McGill questionnaire.
Functional Capacity | From date of randomization (1 week before intervention beginning) up to 5 weeks (T1) and up to 10 weeks (T2; follow-up)
  Functional capacity will be evaluated by Lawton and Brody scale and also by 6 minutes walking test.
Quality of Life | From date of randomization (1 week before intervention beginning) up to 5 weeks (T1) and up to 10 weeks (T2; follow-up)
  Quality of life will be measured through Brazilian version of World Health Organization Quality of Life.
Pulmonary Function | From date of randomization (1 week before intervention beginning) up to 5 weeks (T1) and up to 10 weeks (T2; follow-up)
  This outcome will be assessed through spirometry, assessment of maximal inspiratory pressure and respiratory endurance.
Body Composition | From date of randomization (1 week before intervention beginning) up to 5 weeks (T1) and up to 10 weeks (T2; follow-up)
  Body composition analysis will be carried out by bioelectrical impedance analysis.
Anxiety | From date of randomization (1 week before intervention beginning) up to 5 weeks (T1) and up to 10 weeks (T2; follow-up)
  Anxiety level will be evaluated through Hamilton Anxiety Rating Scale.
Depression | From date of randomization (1 week before intervention beginning) up to 5 weeks (T1) and up to 10 weeks (T2; follow-up)
  Depression will be assessed by Beck's Depression Inventory.
Self-efficacy | Self-efficacy will be assessed after intervention ending.
  Self-efficacy will be evaluated through the Self-efficacy manage chronic disease 6-item scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Paraíba,Department of Psychology, João Pessoa, Paraíba, Brazil